CLINICAL TRIAL: NCT04487886
Title: Duvelisib Ameliorates Manifestations of Pneumonia in Established Novel Coronavirus Infection
Brief Title: Duvelisib Ameliorates Manifestations of Pneumonia in Established Novel Coronavirus Infection (COVID-19)
Acronym: DAMPEN-CI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Verastem, Inc. (Industry)
Responsible Party: Principal Investigator, Edmund Waller, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000701
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — duvelisib

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Duvelisib (Experimental): Participants with severe COVID-19 who do not require mechanical ventilation randomized to receive duvelisib for 14 days.
  Interventions: Drug: Duvelisib
- Placebo (Placebo Comparator): Participants with severe COVID-19 who do not require mechanical ventilation randomized to receive a placebo to match duvelisib for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duvelisib — Duvelisib will be taken orally at an initial dose of 25 milligrams (mg) twice per day for 14 days. The dose will be de-escalated to 15 mg, twice per day, under certain clinical circumstances.
  Other Names: Copiktra
  Arms: Duvelisib
Drug: Placebo — A placebo to match duvelisib will be taken orally twice per day for 14 days.
  Arms: Placebo

SUMMARY:
In this study, patients with severe coronavirus disease 2019 (COVID-19) infection will be randomized to receive duvelisib or a placebo. Participants will be enrolled at Emory University Hospital and will be identified and recruited by their treating physician and research team.

DETAILED DESCRIPTION:
This randomized placebo-controlled phase 2 study will evaluate whether a two-week exposure to duvelisib, a gamma/delta phosphoinositide 3-kinase (PI3K) inhibitor, reduces inflammation in the lungs in patients with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection and COVID-19 who do not require mechanical ventilation at study initiation. The primary objective of the study is to determine the efficacy of duvelisib treatment in preventing death or the need for mechanical ventilation among patients with World Health Organization (WHO)-defined severe COVID-19. Key secondary endpoints will be reductions in oxygen requirements of patients and improvements in their performance status, safety and tolerability of duvelisib in the setting of COVID-19, biomarkers of inflammation, and generation of immunoglobulin G (IgG) and immunoglobulin M (IgM) antibody responses to SARS-Cov-2 spike protein. The study will determine if a two-week exposure to duvelisib beginning soon after presentation with severe COVID-19 warrants further evaluation in a larger clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in participating facility.
* Documentation of pneumonia with radiographic evidence of infiltrates by imaging (e.g., chest x-ray or CT scan).
* Laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other authorized or approved assay in any specimen collected within 72 hours prior to enrollment. Note - An exception must be requested to the Sponsor if ≥72 hours since positive test.
* Symptoms suggestive of severe systemic illness with COVID-19, such as respiratory rate > 30 breaths per minute, heart rate >125 beats per minute, oxygen saturation (O2 sat) in the blood of <93% on room air at sea level or the ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2)< 300
* 18 years of age or older
* Patients with hematological parameters at screening consistent with < grade 2 NCI CTCAE v5.0 toxicity: hemoglobin >8 g/dL, platelet count >50,000 K/mcl, an absolute neutrophil count (ANC) >1,000/mm3, and an absolute lymphocyte count (ALC) >500/mm3.
* Patients with laboratory measurements of liver function at screening consistent with < grade 2 NCI CTCAE v5.0 toxicity: alanine aminotransferase (ALT) < 5 times the upper limit of normal (ULN); aspartate aminotransferase (AST) < 5 times ULN; and bilirubin < 3 times ULN.
* The effects of duvelisib on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) must have a negative serum or urine pr5egnancy test prior to starting therapy. WOCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from enrollment into this study until at least 60 days after the first dose of duvelisib. A woman of childbearing potential (WOCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 2 months after completion of duvelisib administration. WOCBP must have a negative pregnancy test within 24 hours of the first dose of duvelisib.
* The patient must be willing to comply with fertility requirements as below:

  * Total abstinence (when this is in line with the usual practice and lifestyle of the patient) will be accepted. Periodic abstinence (i.e., calendar, ovulation, post-ovulation methods) and withdrawals are not acceptable forms
  * If a female participant is of reproductive potential, the participant (and her partner) must agree to use of one of the following combinations of birth control during the study and for 2 months after the last dose of study drug (or tubal ligation as a single method):

    * Use of a double-barrier method of contraception: condoms (male or female) and a diaphragm or cervical cap with spermicide;
    * Use of an IUD and a barrier method: condoms (male or female, with or without spermicide) or a diaphragm or cervical cap with spermicide;
    * Tubal ligation.
  * Women who are post-menopausal, defined as age greater than 45 and no menses for at least 24 consecutive months, or who have had a hysterectomy, are considered not of reproductive potential.
  * Males must agree to using contraception during the study and for 2 months after the last dose of study drug or have undergone a male sterilization procedure (at least 6 months prior to screening.
  * Use of oral (estrogen and progesterone), injected or implanted hormonal methods of contraception, or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of contraception that comparable efficacy (failure rate <1%). In case of oral contraception, the woman should be stable on the same pill for a minimum of 3 months prior to enrollment on the study.
* Patients must agree not to donate blood, sperm/ova or any other organs while taking protocol therapy and for at least 2 weeks after stopping treatment.
* Willingness and ability of the patient to comply with scheduled visits, drug administration plan, protocol specified laboratory tests, other study procedures and study restrictions
* Evidence of personally signed informed consent indicating that the subject is aware of the life-threatening nature of the disease and has been informed on the procedures to be followed, the experimental nature of the therapy, alternative, potential risks and discomforts, potential benefits and other pertinent aspects of study participation.

Exclusion Criteria:

* Patients requiring mechanical ventilation (intubation or Bi-PAP) at the time randomization.
* Patients receiving any investigational drugs other than drugs or therapies to treat COVID-19, with the exception of investigational immune-modulatory drugs as per section 5.4.
* Pregnant women are excluded from this study because duvelisib is agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with duvelisib, breastfeeding should be discontinued before starting study drug and breastfeeding should not be resumed until at least 1 month after last dose of study drug.
* Clinical suspicion that the etiology of acute illness (acute decompensation) is primarily due to a condition other than COVID-19
* Known contraindication to duvelisib
* Patients with hepatic cirrhosis as defined by symptomatic liver dysfunction; liver fibrosis by biopsy; ALT > 5 times ULN, AST> 5 times ULN, or bilirubin > 3 times ULN.
* Patients with autoimmune diseases or patients on chronic immunosuppressive medications at the time of hospital admission or screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Waller, MD, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The researchers plan to share individual participant data including participant status ordinal score at baseline and end of treatment, study drug allocation, duration of treatment, and survival status at Day 60.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available for sharing at the conclusion of the study and will be available for one year.
Access Criteria: Data will be available for sharing with academic or pharmaceutical investigators for analyses including comparison of DAMPEN-CI results with those from other drug trials in similar patient cohorts. Researchers wishing to use data should email the investigators of DAMPEN-Cl. A summary of the research plan will be required prior to release of the DAMPEN-CI data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Emory University Hospital in Atlanta, Georgia, USA. Participant enrollment began November 18, 2020 and all follow-up assessments were completed by June 10, 2021.
Period: Overall Study
Arm/Group | Duvelisib | Placebo
Started | 25 | 22
Completed | 25 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duvelisib | Placebo | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 15 | 33
  >=65 years | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (12.2) | 58.9 (17.1) | 57.4 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 12 | 29
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Requiring Mechanical Ventilation or Dying
Description: This is a composite endpoint of the number of participants who require mechanical ventilation or who die within four weeks of randomization.
Time Frame: Up to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 22
Participants | 3 | 3

2. Secondary Outcome: Days to Recovery
Description: Time to recovery is measured in days, from the day of randomization to the day of recovery, with recovery defined as a score of equal to or greater than 5 from the eight categories from the National Institute of Allergy and Infectious Diseases (NIAID) ordinal scale. The scale is as follows: 1 = Death, 2 = Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO), 3 = Hospitalized, on non-invasive ventilation or high flow oxygen devices, 4 = Hospitalized, requiring supplemental oxygen, 5 = Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise), 6 = Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care;=, 7 = Not hospitalized, limitation on activities and/or requiring home oxygen, and 8 = Not hospitalized, no limitations on activities.
Time Frame: Up to Day 29
Population: This analysis includes participants who recovered; one participant in the placebo study arm passed away and is not included in this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 21
days | 6.00 (6.19) | 5.29 (4.19)

3. Secondary Outcome: Duration of Hospitalization
Description: The number of days spent hospitalized is presented for both study arms.
Time Frame: Up to Day 29
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 22
days | 6.72 (7.48) | 6.95 (6.41)

4. Secondary Outcome: Days on Study Drug
Description: The number of days that participants took any doses of the study drug that they were randomized to receive is presented for both study arms.
Time Frame: Up to Day 29
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 22
days | 4.6 (3.55) | 5.18 (2.77)

5. Secondary Outcome: Total Doses of Study Drug
Description: The study medication was taken twice per day for 14 days. The number of doses of study medication that was taken is presented for both study arms.
Time Frame: Up to Day 29
Measure: Mean (Standard Deviation); unit: drug doses
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 22
drug doses | 7.76 (6.79) | 8.91 (5.61)

6. Secondary Outcome: Number of Participants Dying
Description: The incidence of death within 29 days of randomization is compared between study arms.
Time Frame: Up to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 22
Participants | 0 | 1

7. Secondary Outcome: Number of Participants Transferred to ICU
Description: The number of participants who were transferred to the intensive care unit (ICU) within 29 days of randomization.
Time Frame: Up to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 22
Participants | 3 | 3

8. Secondary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status Score
Description: The ECOG Performance Status instrument includes a single item assessing overall physical status. Health status is rated on a scale of 0 to 5 where 0 = fully active, 1 = restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, 2 = ambulatory and capable of all selfcare but unable to carry out any work activities, 3 = capable of only limited selfcare, completely disabled, and 5 = dead. Median ECOG performance is compared between study arms.
Time Frame: Between Day 14 and 28, Between Day 29 and 60
Population: This analysis includes participants who were able to be contacted for this assessment, or those with relevant information in the medical chart.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 22 | 22
score on a scale
  Single assessment between Day 14 and 28: number analyzed (Participants) | 22 | 18
  Single assessment between Day 14 and 28 | 2 (1.01) | 1.5 (1.04)
  Single assessment between Day 29 and 60: number analyzed (Participants) | 19 | 22
  Single assessment between Day 29 and 60 | 1 (0.69) | 1 (1.04)

9. Secondary Outcome: Number of Grade III-V Adverse Events
Description: The incidence of grade III-V adverse events or serious adverse events (SAEs), as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 5, is compared between study arms. Grade 3 lab values that required no special treatment are excluded from this outcome measure.
Time Frame: Up to Day 29
Measure: Number; unit: grade III-V adverse events
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 22
grade III-V adverse events | 6 | 3

10. Secondary Outcome: Number of Secondary Bacterial or Viral Infections
Description: The incidence of documented secondary bacterial or viral infections among participants is compared between study arms.
Time Frame: Up to Day 29
Measure: Number; unit: infections
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 22
infections
  Count of bacterial infections | 0 | 1
  Count of viral infections | 0 | 0

11. Secondary Outcome: T Helper 1 (Th1) T Cell Frequency
Description: The mean frequency of Th1 T cells in peripheral blood mononuclear cells (PBMCs) is compared between study arms.
Time Frame: Week 1, Week 2
Measure: Mean (Standard Deviation); unit: percentage of CD4 T cells
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 22
percentage of CD4 T cells
  Week 1 | 19.52 (4.77) | 20.14 (7.52)
  Week 2 | 19.98 (6.24) | 18.27 (6.8)

12. Secondary Outcome: Th17 T Cell Frequency
Description: The mean frequency of Th17 T cells in PBMCs is compared between study arms.
Time Frame: Week 1, Week 2
Measure: Mean (Standard Deviation); unit: percentage of CD4 T cells
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 22
percentage of CD4 T cells
  Week 1 | 2.24 (4.65) | 3.43 (3.78)
  Week 2 | 3.16 (2.44) | 4.25 (3.21)

13. Secondary Outcome: Interleukin-2 (IL-2) Levels
Description: Mean levels of the inflammatory serum biomarker IL-2 is compared between study arms.
Time Frame: Week 1, Week 2
Population: This analysis includes participants who had blood samples obtained at both study time points. Two participants in the placebo arm had samples missing for one of the time points.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 1 | 0.08723 (18.065) | 62.8596 (18.171)
  Week 2 | 17.3632 (40.588) | 0.3158 (32.3258)

14. Secondary Outcome: Interleukin-2 Receptor (IL-2R) Levels
Description: Mean levels of the inflammatory serum biomarker IL-2R is compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 1 | 1172.80 (529.75) | 3569.93 (540.08)
  Week 2 | 912.47 (976.08) | 2005.94 (1207.7)

15. Secondary Outcome: Interleukin-6 (IL-6) Levels
Description: Mean levels of the inflammatory serum biomarker IL-6 is compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 1 | 7.9388 (41.3498) | 149.73 (42.0497)
  Week 2 | 14.2294 (75.829) | 52.2227 (94.026)

16. Secondary Outcome: Interleukin-7 (IL-7) Levels
Description: Mean levels of the inflammatory serum biomarker IL-7 is compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 1 | 4.6018 (54.6831) | 198.80 (55.2375)
  Week 2 | 3.2255 (98.8781) | 48.5118 (123.46)

17. Secondary Outcome: Interleukin-8 (IL-8) Levels
Description: Mean levels of the inflammatory serum biomarker IL-8 is compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 1 | 3.1109 (28.2498) | 104.03 (28.5967)
  Week 2 | 3.4120 (51.3241) | 26.6383 (63.927)

18. Secondary Outcome: Interleukin-10 (IL-10) Levels
Description: Mean levels of the inflammatory serum biomarker IL-10 is compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 1 | 389.02 (838.50) | 808.09 (831.24)
  Week 2 | 658.17 (1411.11) | 250.00 (1836.14)

19. Secondary Outcome: Interferon Gamma-induced Protein 10 (IP-10) Levels
Description: Mean levels of the inflammatory serum biomarker IP-10is compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 1 | 3136.50 (652.84) | 4781.42 (649.35)
  Week 2 | 2956.68 (1122.8) | 3809.83 (1442.4)

20. Secondary Outcome: Macrophage Inflammatory Protein 1alpha (MIP-1a) Levels
Description: Mean levels of the inflammatory serum biomarker MIP-1a is compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 1 | 29.0477 (26.449) | 123.60 (26.8550)
  Week 2 | 43.0115 (48.356) | 57.5810 (60.045)

21. Secondary Outcome: Monocyte Chemoattractant Protein-1 (MCP-1) Levels
Description: Mean levels of the inflammatory serum biomarker MCP-1 are compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 1 | 122.63 (28.2616) | 124.80 (27.9714)
  Week 2 | 255.30 (46.5051) | 187.12 (61.2899)

22. Secondary Outcome: Granulocyte Colony-stimulating Factor (G-CSF) Levels
Description: Mean levels of the inflammatory serum biomarker G-CSF are compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 1 | 8.1585 (42.8679) | 157.86 (43.5125)
  Week 2 | 8.6447 (78.3263) | 39.7275 (97.289)

23. Secondary Outcome: Tumor Necrosis Factor (TNF)-Alpha Levels
Description: Mean levels of the inflammatory serum biomarker TNF-alpha are compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 1 | 1.3291 (21.8406) | 81.0170 (22.236)
  Week 2 | 2.6108 (40.1411) | 17.0332 (49.723)

24. Secondary Outcome: Gene Expression Profile of Regulatory T Cells (Tregs)
Description: Single-cell ribonucleic acid (RNA) sequencing is a powerful gene expression profiling tool to acquire transcriptional level information of each gene. Mean levels of the Tregs will be compared between study arms.
Time Frame: Week 1, Week 2
Population: Due to funding limitations single-cell RNA sequencing was not performed. As the focus of this study was to determine the immune profile consisting of immune cell composition and serum cytokine/chemokine other laboratory experiments provided sufficient data for this purpose.
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Gene Expression Profile of Cluster of Differentiation 8 (CD8)+Interferon Gamma (IFNg)+ Granulocyte-macrophage Colony-stimulating Factor (GM-CSF)+
Description: Single-cell RNA sequencing is a powerful gene expression profiling tool to acquire transcriptional level information of each gene. Mean levels of CD8+IFNg+GM-CSF+ will be compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 24
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Gene Expression Profile of CD8+ T Cell Immunoglobulin and Mucin Domain-containing Protein 3 (Tim3)+ Programmed Cell Death Protein 1 (PD-1)+
Description: Single-cell RNA sequencing is a powerful gene expression profiling tool to acquire transcriptional level information of each gene. Mean levels of CD8+Tim3+PD-1+ will be compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 24
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Gene Expression Profile of Cluster of Differentiation 14 (CD14)+ Cluster of Differentiation (CD16)+ Monocytes
Description: Single-cell RNA sequencing is a powerful gene expression profiling tool to acquire transcriptional level information of each gene. Mean levels of CD14+CD16+ monocytes will be compared between study arms.
Time Frame: Week 1, Week 2
Population: as for outcome 24
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Immunoglobin G (IgG) Antibodies
Description: Median titers of IgG antibodies to SARS-CoV-2 at 4 weeks will be assessed for both study arms.
Time Frame: Week 4
Population: Due to budget limitations other laboratory experiments were prioritized and Immunoglobulin G (IgG) antibodies were not measured.
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Number of Participants Surviving
Description: Overall survival is defined as days from randomization to death and censored at last follow up.
Time Frame: Up to Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 25 | 22
Participants | 25 | 21

30. Other Pre Specified Outcome: Vasoactive Intestinal Peptide (VIP)
Description: VIP is a peptide hormone with immunosuppressive properties. Mean levels VIP will be compared between study arms.
Time Frame: Week 1, Week 2
Population: Due to budget limitations other laboratory experiments were prioritized and VIP (an exploratory outcome) was not analyzed.
Arm/Group | Duvelisib | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time study treatment began until 14 days following cessation of duvelisib or placebo (up to Day 29). Survival status was assessed up to Day 60.
Description: Adverse events that began or worsened after informed consent to participate was given were recorded.
Arm/Group | Duvelisib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/22
Serious Adverse Events (participants affected / at risk) | 6/25 | 2/22
Other Adverse Events (participants affected / at risk) | 5/25 | 5/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib (N=25) | Placebo (N=22)
Transfer to ICU and/or initiation of mechanical ventilation (General disorders) | 3 | 2
Post-discharge hospitalization (General disorders) | 3 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib (N=25) | Placebo (N=22)
High alanine transaminase (ALT) - grade 2 (Hepatobiliary disorders) | 0 | 1
Leukopenia - grade 2 (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia - grade 2 or 3 (Blood and lymphatic system disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT04487886/Prot_SAP_000.pdf